CLINICAL TRIAL: NCT05193435
Title: Comparison of Stabilization Exercises and Pelvic Floor Muscle Training in Women With Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/01/2
Record Dates: First submitted 2022-01-02; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor exercise group (Experimental): Pelvic floor exercises for muscle fiber types I and II will performed 3 days a week for 8 weeks
  Interventions: Other: Pelvic floor exercises
- Stabilization exercise group (Active Comparator): Lumbar spinal stabilization exercises will performed 3 days a week for 8 weeks
  Interventions: Other: Stabilization exercises

INTERVENTIONS:
Other: Pelvic floor exercises — Pelvic floor exercises for types I and II muscle fibers will be performed
  Arms: Pelvic floor exercise group
Other: Stabilization exercises — Lumbar spinal stabilization exercises will be performed
  Arms: Stabilization exercise group

SUMMARY:
The aim of the study was to compare the effects of stabilization exercises and pelvic floor muscle training in women with stress urinary incontinence.

DETAILED DESCRIPTION:
Stress urinary incontinence is involuntary urinary incontinence with increased intraabdominal pressure. Different exercise approaches such as pelvic floor exercises and stabilization exercises are used in these patients. There is a need for studies comparing the effects of these exercises.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-65 who have symptoms of stress or stress-dominant mixed urinary incontinence, who volunteered to participate in the study

Exclusion Criteria:

* Those who are pregnant, have communication and cooperation problems, have a concomitant neurological or rheumatological disease, have a history of surgery involving the abdominal and pelvic regions in the last year, have undergone spine surgery, those diagnosed with pure urge urinary incontinence or mixed type incontinence, those with advanced pelvic organ prolapse, those with a spinal deformity (such as scoliosis), the presence of orthopedic problems in the lower extremities (such as lower extremity shortness, presence of deformity etc.) and vestibular system disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence severity | change from baseline at 8 weeks
  Urinary incontinence severity will be measured with A 1-hour pad test

SECONDARY OUTCOMES:
Urinary symptoms | change from baseline at 8 weeks
  Urinary symptoms will be evaluated with International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form
Life quality | change from baseline at 8 weeks
  Life quality will be assessed with King's Health Questionnaire.
Pelvic floor muscle activation response | change from baseline at 8 weeks
  Pelvic floor muscle activation response will be measured with a portable EMG-Biofeedback device.
Pelvic floor muscle strength | change from baseline at 8 weeks
  Pelvic floor muscle strength will be evaluated with Modified Oxford Scale
Core stability | change from baseline at 8 weeks
  Core stability will be evaluated with Sahrmann Test using the pressure stabilizer.
Balance | change from baseline at 8 weeks
  Balance will be evaluated with Biodex Balance System as static and dynamic
Spinal function | change from baseline at 8 weeks
  Spinal function will be evaluated with the Spinal Mouse device in standing position.
Subjective perception of improvement | After treatment (at 8 week)
  Subjective perception of improvement will be measured with a four-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322